CLINICAL TRIAL: NCT00292396
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Safety and Efficacy of Subcutaneous Injections of ABT-874 vs. Placebo in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety of ABT-874 in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M05-736
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Active Comparator): Anti IL-12 monoclonal antibody/ABT-874, up to 12 weeks, 200 mg every week for 12 weeks
  Interventions: Drug: Anti IL-12 monoclonal antibody/ABT-874
- 2 (Active Comparator): Anti IL-12 monoclonal antibody/ABT-874, 200 mg QOW for 12 weeks
  Interventions: Drug: Anti IL-12 monoclonal antibody/ABT-874
- 3 (Active Comparator): Anti IL-12 monoclonal antibody/ABT-874, 100 mg QOW in 12 weeks
  Interventions: Drug: Anti IL-12 monoclonal antibody/ABT-874
- 4 (Active Comparator): Anti IL-12 monoclonal antibody/ABT-874, 200 mg times 4 doses in 12 weeks
  Interventions: Drug: Anti IL-12 monoclonal antibody/ABT-874
- 5 (Active Comparator): Anti IL-12 monoclonal antibody/ABT-874, 200 mg times 1 dose in 12 weeks
  Interventions: Drug: Anti IL-12 monoclonal antibody/ABT-874
- 6 (Placebo Comparator): placebo, 12 doses
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Anti IL-12 monoclonal antibody/ABT-874 — Please see Arm Description for intervention description and details.
  Arms: 1; 2; 3; 4; 5
Drug: placebo — 12 doses
  Arms: 6

SUMMARY:
The purpose of the study is to assess the safety and efficacy of ABT-874 in the treatment of moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject was age 18 or older and in good health (Investigator discretion) with a recent stable medical history.
* Subject had a clinical diagnosis of psoriasis for at least 6 months, and had moderate to severe plaque psoriasis

Exclusion Criteria:

* Subject had previously received systemic or biologic anti-IL-12 therapy
* Subject cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot avoid UVB or PUVA phototherapy
* Subject is taking or requires oral or injectable corticosteroids
* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with clinical response relative to Baseline PASI score | Week 12, Week 40 and Week 60

SECONDARY OUTCOMES:
Quality of Life Surveys | Week 12, Week 48 and Week 60
Clinical response indicators | Week 12, Week 48 and Week 60
Safety parameters | Monthly through duration of study
PGA Assessment | Week 12, Week 40 and Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaul, MD, Study Chair — AbbVie
Locations (24):
- United States (16):
  - Site Reference ID/Investigator# 3351, San Diego, California
  - Site Reference ID/Investigator# 3347, Alpharetta, Georgia
  - Site Reference ID/Investigator# 3348, Skokie, Illinois
  - Site Reference ID/Investigator# 993, Indianapolis, Indiana
  - Site Reference ID/Investigator# 990, Boston, Massachusetts
  - Site Reference ID/Investigator# 3349, St Louis, Missouri
  - Site Reference ID/Investigator# 992, Cincinnati, Ohio
  - Site Reference ID/Investigator# 991, Lake Oswego, Oregon
  - Site Reference ID/Investigator# 3367, Portland, Oregon
  - Site Reference ID/Investigator# 3346, Johnston, Rhode Island
  - Site Reference ID/Investigator# 994, Nashville, Tennessee
  - Site Reference ID/Investigator# 3350, Dallas, Texas
  - Site Reference ID/Investigator# 796, Houston, Texas
  - Site Reference ID/Investigator# 2081, Salt Lake City, Utah
  - Site Reference ID/Investigator# 3366, Norfolk, Virginia
  - Site Reference ID/Investigator# 989, Seattle, Washington
- Canada (8):
  - Site Reference ID/Investigator# 3361, Halifax
  - Site Reference ID/Investigator# 985, Laval
  - Site Reference ID/Investigator# 987, London
  - Site Reference ID/Investigator# 3364, Montreal
  - Site Reference ID/Investigator# 794, North Bay
  - Site Reference ID/Investigator# 988, Québec
  - Site Reference ID/Investigator# 795, Waterloo
  - Site Reference ID/Investigator# 3360, Windsor

REFERENCES:
- [Derived] Kimball AB, Gordon KB, Langley RG, Menter A, Chartash EK, Valdes J; ABT-874 Psoriasis Study Investigators. Safety and efficacy of ABT-874, a fully human interleukin 12/23 monoclonal antibody, in the treatment of moderate to severe chronic plaque psoriasis: results of a randomized, placebo-controlled, phase 2 trial. Arch Dermatol. 2008 Feb;144(2):200-7. doi: 10.1001/archdermatol.2007.63. PMID 18283176